CLINICAL TRIAL: NCT04786574
Title: A Phase 3b Multicenter Open-label Trial of the Safety, Tolerability, and Efficacy of Tolvaptan in Infants and Children 28 Days to Less Than 12 Weeks of Age With Autosomal Recessive Polycystic Kidney Disease (ARPKD)
Brief Title: A Study to See if Tolvaptan Can Delay Dialysis in Infants and Children Who at Enrollment Are 28 Days to Less Than 12 Weeks Old With Autosomal Recessive Polycystic Kidney Disease (ARPKD)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped before enrolling any participants.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-12-204
Record Dates: First submitted 2021-02-19; First posted 2021-03-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Autosomal Recessive Polycystic Kidney Disease (ARPKD)
Keywords: ARPKD; Tolvaptan; Polycystic Kidney Disease; Autosomal Recessive Polycystic Kidney Disease; Renal Cysts; Nephromegaly; Oligohydramnios; Anhydramnios
MeSH Terms: conditions — Polycystic Kidney, Autosomal Recessive; Polycystic Kidney Diseases; Oligohydramnios | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tolvaptan (OPC-41061) (Experimental)
  Interventions: Drug: Tolvaptan (OPC-41061)

INTERVENTIONS:
Drug: Tolvaptan (OPC-41061) — Tolvaptan suspension will be administered orally or via nasogastric tube at doses of 0.15 mg/kg once daily in the AM, 0.30 mg/kg once daily in the AM, 0.5 mg/kg once daily in the AM, 0.75 mg/kg split dose (0.5 mg/kg AM and 0.25 mg/kg 8 hours later), and 1 mg/kg split dose (0.67 mg/kg AM and 0.33 mg/kg 8 hours later) based on age. Treatment duration is 2 years.

SUMMARY:
The primary objective of this study is to evaluate the effect of tolvaptan on the need for renal replacement therapy in pediatric subjects with autosomal recessive polycystic kidney disease (ARPKD)

DETAILED DESCRIPTION:
Tolvaptan has been demonstrated to delay the decline of kidney function in adults with rapidly progressing ADPKD (CKD stages 1 to 3), a closely related indication to ARPKD, as measured by estimated glomerular filtration rate (eGFR) and Total Kidney Volume (TKV).

The trial will be the first trial of tolvaptan in a pediatric ARPKD population.

Participants in this study will be assigned to tolvaptan for 24 months and closely monitored over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 28 days and < 12 weeks of age, inclusive at the time of enrollment.
2. Must have clinical and imaging features that are consistent with a diagnosis of ARPKD with all the following characteristics:

   * Nephromegaly (> 2 standard deviations from age-appropriate standard via ultrasound)
   * Multiple renal cysts
   * History of oligohydramnios or anhydramnios
3. Ability for parent or guardian to provide written, informed consent prior to initiation of any trial-related procedures, and ability, in the opinion of the principal investigator, to comply with all the requirements of the trial.

Exclusion Criteria:

1. Premature birth (≤ 32 weeks gestational age)
2. Anuria or RRT, defined as intermittent or continuous hemodialysis, peritoneal dialysis, hemofiltration, hemodiafiltration or history of kidney transplantation
3. Evidence of syndromic conditions associated with renal cysts (other than ARPKD)
4. Abnormal liver function tests including ALT and AST, > 1.2 × ULN
5. Parents with renal cystic disease
6. Need for chronic diuretic use
7. Cannot be monitored for fluid balance
8. Has or at risk of having sodium and potassium electrolyte imbalances
9. Has or at risk of having significant hypovolemia as determined by investigator
10. Clinically significant anemia, as determined by investigator
11. Severe systolic dysfunction defined as ejection fraction < 14%
12. Serum sodium levels < 130 mmol/L or >145 mmol/L
13. Taking any other experimental medications
14. Require ventilator support
15. Taking medications known to induce CYP3A4
16. Having an infection including viral that would require therapy disruptive to IMP dosing
17. Platelet count <50,000 µL
18. Significant Portal Hypertension
19. Bladder dysfunction or difficulty voiding
20. Taking vasopressin agonist
21. Having concomitant illness or taking medications that are likely to confound endpoint assessments.
22. History of cholangitis
23. Received or scheduled to receive a liver transplant

Ages: 4 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects that will have Renal Replacement Therapy (RRT) by 1 year of age. | From Enrollment to 1 year of age

SECONDARY OUTCOMES:
Rate of change of eGFR by Schwartz formula from pre-treatment to after 2 years of treatment | From Enrollment to 2 years of age
Palatability of the suspension formulation as assessed by a parent questionnaire immediately after and within 15-20 minutes after the first oral dose | From Enrollment to 2 years of age
Acceptance of the suspension formulation as assessed by a parent questionnaire immediately after and within 15-20 minutes after the first oral dose | From Enrollment to 2 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Olga Sergeyeva, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.

IPD SHARING:
Plan to Share IPD: No